CLINICAL TRIAL: NCT05001555
Title: Efficacy and Safety of the Combination Dexketoprofen / Vitamin B Vs Dexketoprofen in the Treatment of Pain in Patients with Post-traumatic Cervical Sprain Grade I-II of the Quebec Scale.
Brief Title: Efficacy and Safety of Dexketoprofen/Vitamin B Vs Dexketoprofen for Post-traumatic Cervical Sprain Grade I-II
Acronym: WHIPLASH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIL-30242-III-20 (1)
Record Dates: First submitted 2021-07-29; First posted 2021-08-12 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Acute Low Back Pain
MeSH Terms: interventions — dexketoprofen trometamol; Folic Acid; Fumigant 93

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Dexketoprofen/Vitamin B (Thiamine mononitrate/Pyridoxine hydrochloride/Cyanocobalamin) (Experimental): Group A:
  Dexketoprofen/Vitamin B (Thiamine mononitrate/Pyridoxine hydrochloride/Cyanocobalamin), 1 capsule, orally, every 8 hours, for 7 days.
  Interventions: Drug: Dexketoprofen/Vitamin B
- Group B: Dexketoprofen (Active Comparator): Group B: Dexketoprofen, 1 tablet, orally, every 8 hours, for 7 days.
  Interventions: Drug: Dexketoprofen

INTERVENTIONS:
Drug: Dexketoprofen/Vitamin B — 1 capsule containing 25 mg of dexketoprofen / vitamin B (thiamine mononitrate 100 mg, Pyridoxine hydrochloride 50 mg, Cyanocobalamin 0.50 mg), orally, every 8 hours, for 7 days.
  Other Names: D/VitB
  Arms: Group A: Dexketoprofen/Vitamin B (Thiamine mononitrate/Pyridoxine hydrochloride/Cyanocobalamin)
Drug: Dexketoprofen — 1 tablet of dexketoprofen 25 mg, orally, every 8 hours, for 7 days.
  Other Names: D
  Arms: Group B: Dexketoprofen

SUMMARY:
Phase IIIb, multicenter, prospective, randomized, double-blind study to evaluate the fixed combination of Desketoprofen / Vitamin B in the management of acute pain in patients with cervical sprain grade I-II of the Quebec scale.

DETAILED DESCRIPTION:
Study to evaluate the efficacy and safety of the Dexketoprofen / Vitamin B combination versus dexketoprofen for the management of acute pain secondary to post-traumatic cervical sprain grade I-II of the Quebec scale, evaluated by means of the Visual Analogue Scale (VAS). To compare the degree of disability due to neck pain measured through the Northwick Park Neck Pain Questionnaire in Spanish version on days 3, 5, and 7 compare to its baseline measurement between the treatment groups. Compare the proportion of subjects requiring rescue medication during the study between treatment groups. Describe the frequency and intensity of adverse events presented during the study.

ELIGIBILITY:
Inclusion Criteria:

* Any sex.
* That the subject agree to participate in the study and give your written informed consent.
* Age> 18 years old at the beginning of the study.
* Diagnosis of a grade I or Grade II cervical sprain on the Quebec scale of no more than 3 days.
* Visual Analog Scale (VAS) ≥4 cm.
* Women of childbearing potential using a contraceptive method (barrier, oral hormonal, injectable, subdermal), menopausal or surgically sterile.

Exclusion Criteria:

* Patient in whom the drug is contraindicated for medical reasons.
* History of allergic reaction to NSAIDs, thiamine, pyridoxine and cyanocobalamin or hypersensitivity to the components of the formula.
* A significant history of gastrointestinal disorders (for example: Gastric Ulcer, Crohn's Disease, Ulcerative Colitis, etc.)
* Previous treatment with opioids reported in the medical history.
* History of inflammatory arthritis (eg rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, gout).
* History of chronic pain (eg, fibromyalgia), metastasis, and Paget's disease.
* History of alcohol or drug abuse in the last year according to DSM-V.
* Clinical and radiological data of cervical sprain grade III or IV of the Quebec scale.
* History of illness or injury for more than 6 months in the neck or cervical spine
* Patient with symptoms of spinal cord injury (weakness, incoordination or paralysis in any part of the body, numbness, tingling or loss of sensation in the hands, fingers, feet or toes, etc.)
* History of severe acute or chronic liver failure.
* History of moderate to severe renal failure.
* A significant history of coagulation problems (Von Willembrand, hemophilia, vitamin K deficiency, etc.).
* At medical discretion, a disease that affects the prognosis and prevents outpatient management, for example, but not restricted to: end-stage cancer, kidney, heart, respiratory or liver failure or mental illness or with scheduled surgical or hospital procedures.
* History / presence of any disease or condition that, in the opinion of the Investigator, could pose a risk to the patient or confuse the efficacy and safety of the study results.
* Oncological patients (except basal cell skin cancer) or with serious diseases that, in the opinion of the investigator, have a serious prognosis or a life expectancy of less than 1 year, as well as mental illnesses.
* Patients with symptoms suggesting an active COVID-19 infection (ie, fever, cough, dyspnea) and / or contact in the past 14 days with a suspected or positive COVID-19 patient.
* Patient is participating in another clinical study involving an investigational treatment or participated in one in the previous 4 weeks.
* Patients whose participation in the study may be influenced (employment relationship with the research center or sponsor, inmates, etc.)
* Positive pregnancy test, women who are pregnant, breastfeeding or planning a pregnancy while conducting the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Changes in pain intensity | Baseline, 3, 5 and 7 days
  Compare changes in pain intensity measured by the visual analog scale (VAS) between treatment groups. The VAS for pain is a straight line of 10 centimeters in which one end means no pain and the other end means the worst pain imaginable.
Change in the degree of disability | Baseline, 3, 5 and 7 days
  Compare the degree of disability due to neck pain measured through the Northwick Park Neck Pain Questionnaire Spanish version between the treatment groups. It includes 9 questions or items (intensity of neck pain, and sleep, pins and needles in the arms at night, duration of symptoms, lifting weights, reading and watching TV, work, social activities and driving). Each of these questions has five possible answers with a score of 0 to 4, from less to greater intensity and severity respectively.
Proportion of subjects requiring rescue medication | 7 days
  Compare the proportion of subjects requiring rescue medication during the study between treatment groups.
Adverse events frequency | 7 days
  Compare the proportion of subjects that presented an adverse event between treatment groups.
Adverse events intensity | 7 days
  Compare the intensity of adverse events presented during the study, between treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Delgado García, M.D, Principal Investigator — IMACEN S.A. de C.V.,; Adelfia Urenda Quezada, M.D, Principal Investigator — Mediadvance Clinical S.A.P.I. de C.V.; Ma. Dolores Alonso Martínez, M.D, Principal Investigator — CICMEX Centro de Investigación Clínica de México; Juan B Alcocer Herrera, M.D, Principal Investigator — INBIOMEDyC Querétaro
Locations (1):
- Laboratorio Silanes, S.A. de C.V., Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spitzer WO, Skovron ML, Salmi LR, Cassidy JD, Duranceau J, Suissa S, Zeiss E. Scientific monograph of the Quebec Task Force on Whiplash-Associated Disorders: redefining "whiplash" and its management. Spine (Phila Pa 1976). 1995 Apr 15;20(8 Suppl):1S-73S. No abstract available. PMID 7604354
- [Background] Rodriquez AA, Barr KP, Burns SP. Whiplash: pathophysiology, diagnosis, treatment, and prognosis. Muscle Nerve. 2004 Jun;29(6):768-81. doi: 10.1002/mus.20060. PMID 15170609
- [Background] Hartling L, Brison RJ, Ardern C, Pickett W. Prognostic value of the Quebec Classification of Whiplash-Associated Disorders. Spine (Phila Pa 1976). 2001 Jan 1;26(1):36-41. doi: 10.1097/00007632-200101010-00008. PMID 11148643
- [Background] Bagan JV, Lopez Arranz JS, Valencia E, Santamaria J, Eguidazu I, Horas M, Forns M, Zapata A, Artigas R, Mauleon D. Clinical Comparison of Dexketoprofen Trometamol and Dipyrone in Postoperative Dental Pain. J Clin Pharmacol. 1998 Dec;38(S1):55S-64S. doi: 10.1002/jcph.1998.38.s1.55. PMID 29023870
- [Background] Ponce-Monter HA, Ortiz MI, Garza-Hernandez AF, Monroy-Maya R, Soto-Rios M, Carrillo-Alarcon L, Reyes-Garcia G, Fernandez-Martinez E. Effect of diclofenac with B vitamins on the treatment of acute pain originated by lower-limb fracture and surgery. Pain Res Treat. 2012;2012:104782. doi: 10.1155/2012/104782. Epub 2011 Oct 31. PMID 22135737
- [Background] Curatolo M, Sveticic G. Drug combinations in pain treatment: a review of the published evidence and a method for finding the optimal combination. Best Pract Res Clin Anaesthesiol. 2002 Dec;16(4):507-19. doi: 10.1053/bean.2002.0254. PMID 12516888
- [Background] Levin OS, Moseikin IA. [Vitamin B complex (milgamma) in the treatment of vertebrogenic lumbosacral radiculopathy]. Zh Nevrol Psikhiatr Im S S Korsakova. 2009;109(10):30-5. Russian. PMID 20037567
- [Background] Kuhlwein A, Meyer HJ, Koehler CO. [Reduced diclofenac administration by B vitamins: results of a randomized double-blind study with reduced daily doses of diclofenac (75 mg diclofenac versus 75 mg diclofenac plus B vitamins) in acute lumbar vertebral syndromes]. Klin Wochenschr. 1990 Jan 19;68(2):107-15. doi: 10.1007/BF01646857. German. PMID 2138683
- [Background] Perez-Flores E, Medina-Santillan R, Reyes-Garcia G, Mateos-Garcia E. Combination of diclofenac plus B vitamins in acute pain after tonsillectomy: a pilot study. Proc West Pharmacol Soc. 2003;46:88-90. No abstract available. PMID 14699896
- [Background] Mibielli MA, Geller M, Cohen JC, Goldberg SG, Cohen MT, Nunes CP, Oliveira LB, da Fonseca AS. Diclofenac plus B vitamins versus diclofenac monotherapy in lumbago: the DOLOR study. Curr Med Res Opin. 2009 Nov;25(11):2589-99. doi: 10.3111/13696990903246911. PMID 19731994
- [Background] Gonzalez T, Balsa A, Sainz de Murieta J, Zamorano E, Gonzalez I, Martin-Mola E. Spanish version of the Northwick Park Neck Pain Questionnaire: reliability and validity. Clin Exp Rheumatol. 2001 Jan-Feb;19(1):41-6. PMID 11247324
- [Background] Gaskell H, Derry S, Wiffen PJ, Moore RA. Single dose oral ketoprofen or dexketoprofen for acute postoperative pain in adults. Cochrane Database Syst Rev. 2017 May 25;5(5):CD007355. doi: 10.1002/14651858.CD007355.pub3. PMID 28540716
- [Derived] Delgado-Garcia P, Alcocer-Herrera JB, Urenda-Quezada A, Alonso-Martinez MD, Bautista-Mendoza MA, Romero-Antonio Y, Mora-Villalobos JC, Sander-Padilla JG, Rios-Brito KF, Rodriguez-Vazquez IC, Gonzalez-Canudas J. A Randomized Control Trial of Dexketoprofen/Vitamin B (Thiamine, Pyridoxine and Cyanocobalamin) Fixed-Dose Combination in Post-Traumatic Grade I-II Cervical Sprains. Clin Drug Investig. 2024 Jun;44(6):413-424. doi: 10.1007/s40261-024-01370-2. Epub 2024 Jun 6. PMID 38842764